CLINICAL TRIAL: NCT02637349
Title: Polaris Oncology Survivor Transition (POST) System
Acronym: POST
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Polaris Health Directions (Industry)
Collaborators: University of Massachusetts, Worcester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2R42CA174048-03 (NIH)
Record Dates: First submitted 2015-12-16; First posted 2015-12-22 (Estimated); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Aftercare

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- POST SCP (Experimental): Patient receives Survivorship Care Plan (SCP) after active treatment ends. It will be discussed with the patient. SCP includes medical and psychosocial history, medical contact information, 5-year follow-up plan and educational materials.
  Interventions: Behavioral: POST Intervention
- POST TAU (Active Comparator): Patient receives treatment as usual (TAU) after active treatment ends.
  Interventions: Behavioral: POST Treatment as Usual

INTERVENTIONS:
Behavioral: POST Intervention — POST Intervention group will receive a tailored survivorship care plan (SCP) at the end of their active treatment. The SCP will be discussed with them. Patient will be asked about satisfaction with the end of treatment session.
  Arms: POST SCP
Behavioral: POST Treatment as Usual — The POST control group may receive a survivorship care plan (SCP) as part of treatment as usual though it is not a usual procedure. They will be asked about their satisfaction with the end of treatment session.
  Arms: POST TAU

SUMMARY:
The POST's public health impact is likely to be substantial because it will improve cancer survivorship planning, which is currently an important deficiency in cancer care recognized by the Institute of Medicine and the American College of Surgeons.

The POST may have many potential benefits for patients such as:

1. improved long-term health outcomes;
2. improved psychosocial outcomes and quality of life;
3. smoother transitions back into old and new life roles; and
4. improved continuity and coordination of care between providers.

Most importantly, the POST's influence may reach beyond the patients it directly serves as it could help scientists and health care providers understand the potential benefits of cancer survivorship planning and how to best design and implement survivorship planning when patients are ending treatment for cancer.

DETAILED DESCRIPTION:
By January 2015, oncology care providers will be expected to craft Survivorship Care Plans (SCPs) for all individuals ending active treatment for cancer; however, there is a lack of systematic study of the impact survivorship planning has on patients, providers, or healthcare systems. The Polaris Oncology Survivorship Transition (POST) program is a web-based system that incorporates recommendations from the Institute of Medicine (IOM) and American College of Surgeons (ACS) to assist with cancer survivorship planning. It is a patient-centered approach that integrates input from both the treating oncology team and the patient. Phase 1 built and iteratively modified (N=25) the POST system and Phase 2 will test whether the SCPs impact patient and provider outcomes using a single blind, randomized controlled trial (RCT). Breast cancer patients (n=230) transitioning out of active treatment will be recruited and randomly assigned to receive Treatment as Usual (n=115) or the POST (n=115). All participants will be assessed at 1, 3, and 6 months by a research assistant blind to baseline status and group assignment. Primary outcomes will include quality of life, mechanisms of action such as confidence in entering survivorship, and other outcomes such as (1) depression and anxiety, (2) adherence to medical and behavioral health recommendations, (3) health care utilization, and (4) patient and provider satisfaction with the POST system.The POST will innovate the clinical setting through being the first system to produce computer generated tailored survivorship plans fully reflecting IOM recommendations and the new ACS 2015 requirements; incorporating information from both the oncology provider and the patient; featuring readily available "plug in" for two-way electronic health record integration; providing dynamic, electronic referrals for specialized support services; and facilitating care coordination between the oncologist and PCP. This study's impact will be significant. If hypotheses are confirmed, clear scientific evidence will exist for supporting survivorship care planning into oncology clinical practice. If hypotheses are disconfirmed, important lessons will guide future directions for care planning, including whether failure to affect outcomes was due to failure to impact several hypothesized mechanisms of action.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Confirmed diagnosis of breast cancer (not metastatic)
* A final active treatment appointment scheduled with oncology team
* Able to read or understand English at a 6th grade level

Exclusion Criteria:

* Altered mental status (e.g., psychosis, delirium, disorientation)
* Visual problems preventing them from reading the assessment and reports
* Severe illness that would preclude conversation or interface with a computer (e.g.,persistent nausea/vomiting, severe pain)
* Unable to read or understand English at a 6th grade level
* Characteristics that would prevent adequate follow-up (e.g., lack of a telephone)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2016-11-30 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Changes in Quality of Life | 1,3, 6 months after entering the study
  Quality of life will be measured at baseline and at the follow-ups using the City of Hope Quality of Life measure. Improvement in quality of life is the primary goal of survivorship planning.

SECONDARY OUTCOMES:
Changes in Confidence in Transitioning to Survivorship | 1,3,6 months after entering the study
  National Cancer Institute (NCI) and the Institute of Medicine (IOM) have emphasized that SCPs should help improve patients' feelings of preparedness and confidence in managing and understanding the next steps at the end of treatment. This will be measured at baseline and follow-up sessions using the Confidence in Survivorship Information Questionnaire (CSI).
Changes in Depression | 1,3,6 months after entering study
  Changes in depression will be measured by the Patient Health Questionnaire -9 (PHQ-9).
Changes in Anxiety | 1,3,6 months after entering study
  Changes in anxiety will be measured by the General Anxiety Disorder 7-item measure (GAD-7).
Change in Health care utilization | 6-months after entering the study
  Participants' medical charts will be reviewed six months after termination of active treatment for frequency and appropriateness of oncology, primary care, and emergency room visits, as well as hospitalizations.
Change in Patient Satisfaction and Usefulness of SCP | 1,3,6 months after entering the study
  Patients will be asked to assess their satisfaction with the POST program and with the content and quality of the SCP.
Change in Patient Satisfaction with the POST system | 1,3,6 months after entering the study
  Patients will be asked to assess their satisfaction with the POST system.
Change in Provider Satisfaction with the POST system | 1,3,6 months after entering the study
  Providers will be asked to assess their satisfaction with the POST system.

CONTACTS AND LOCATIONS:
Overall Officials: Erin O'Hea, PhD, Principal Investigator — University of Massachusetts, Worcester
Locations (1):
- University of Massachusetts Medical School-Cancer Center, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] O'Hea EL, Creamer S, Flahive JM, Keating BA, Crocker CR, Williamson SR, Edmiston KL, Harralson T, Boudreaux ED. Survivorship care planning, quality of life, and confidence to transition to survivorship: A randomized controlled trial with women ending treatment for breast cancer. J Psychosoc Oncol. 2022;40(5):574-594. doi: 10.1080/07347332.2021.1936336. Epub 2021 Jun 20. PMID 34151734